CLINICAL TRIAL: NCT04636515
Title: A Phase 2, Open-label, Single-arm，Multicenter Study of F520 in Patients With Urothelial Carcinoma
Brief Title: A Phase Ⅱ Study of F520 in Patients With Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-006
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Locally Advanced or Metastatic Urothelial Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: F520

INTERVENTIONS:
Drug: F520 — 200mg，Q3W

SUMMARY:
This is a multicenter, Phase 2 study to evaluate the efficacy and safety of the anti- programmed cell death-1(PD-1) monoclonal antibody F520 in participants with locally advanced or metastatic Urothelial Cancer (UC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed,locally advanced（T4b,any N or any T,N2-3 or metastatic carcinoma（including renal pelvic, ureter bladder and urethra）;
2. Cohort 1：Patients with First-line platinum ineligible must meet criteria for either option a or option b (below):

   1. Has a tumor(s) with PD-L1 combined positive and is considered ineligible to receive cisplatin-based combination therapy, based on 1 of the following:

      * Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 2 within 7 days prior to randomization
      * National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade ≥2 audiometric hearing loss
      * NCI CTCAE Version 5.0 Grade ≥2 peripheral neuropathy OR
   2. In the opinion of the investigator, is considered ineligible to receive any platinum-based chemotherapy (i.e., ineligible for cisplatin and carboplatin) based on:

      * ECOG PS of 2 within 7 days prior to randomization. and ≥1 of the following:
      * Documented visceral metastatic disease
      * NCI CTCAE Version 5.0 Grade ≥2 audiometric hearing loss
      * NCI CTCAE Version 5.0 Grade ≥2 peripheral neuropathy

Cohort 2: Inoperable Patients in sencond line（or beyond）with locally advanced or metastatic urothelial carcinoma who have disease recurrence or progression during or after a platinum-based chemotherapy regimen;

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
* Calculated creatinine clearance ≥ 30 milliliter (mL)/min (Cockcroft-Gault formula)

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1 agent or with CTLA-4 receptor;
2. Has a known hypersensitivity to anti-PD-1 / PD-L1 agent;
3. Known pia meningeal metastasis or active central nervous system (CNS) metastasis revealed by CT or MRI. Participants with asymptomatic brain metastases may participate without evidence of progression for at least 1 month.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the investigator | Approximately 24 months
  ORR is defined as CR+PR